CLINICAL TRIAL: NCT06747767
Title: Early Outcomes of Arthroscopic Versus Open Reduction for Developmental Dysplasia of the Hip in Children: A Randomized Controlled Trial
Brief Title: Early Outcomes of Arthroscopic Versus Open Reduction for Developmental Dysplasia of the Hip in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Abdulkadr Muhammed S. Alany, University Faculty, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Developmental Dysplasia of the Hip (DDH)
Keywords: Arthroscopic-assisted reduction; Developmental dysplasia of the hip; Open surgical reduction; Pediatric orthopedic surgery; Avascular necrosis
MeSH Terms: conditions — Developmental Dysplasia of the Hip; Osteonecrosis | interventions — Arthroscopy; Open Fracture Reduction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopy (Experimental): Arthroscopic Reduction for Developmental Dysplasia of the Hip in Children
  Interventions: Procedure: Arthroscopy
- Open Reduction (Experimental): Open Reduction for Developmental Dysplasia of the Hip in children
  Interventions: Procedure: Open reduction

INTERVENTIONS:
Procedure: Arthroscopy — Arthroscopy
  Arms: Arthroscopy
Procedure: Open reduction — Open reduction
  Arms: Open Reduction

SUMMARY:
This study was designed to determine whether arthroscopic-assisted reduction offers better early surgical outcomes than open reduction for treating developmental dysplasia of the hip in children. By comparing these two approaches, the researchers sought to find out if using an arthroscopic-assisted method could lower redislocation rates, shorten operative time, reduce blood loss, maintain acceptable acetabular alignment, and potentially decrease the risk of complications such as avascular necrosis, thereby improving the quality of care and long-term hip function for affected children.

DETAILED DESCRIPTION:
This investigation evaluates two distinct surgical strategies for managing developmental dysplasia of the hip (DDH) in young children using a comparative, parallel-group design. The technical approach under consideration involves an arthroscopic-assisted procedure, which provides direct visualization of the hip joint structures through minimally invasive portals. By employing specialized instruments and an arthroscopic camera system, surgeons can assess ligamentous and capsular integrity, identify obstacles to proper femoral head positioning, and address intra-articular pathologies with potentially less disruption to the vascular supply and surrounding soft tissues than is typical in conventional open surgery. The surgical team implemented stringent measures to maintain uniformity in anesthesia protocols, operative setup, and postoperative immobilization strategies, ensuring that any observed differences would more likely be attributable to the surgical technique rather than confounding variables. Additionally, advanced imaging modalities, including fluoroscopic guidance where appropriate, were used intraoperatively to confirm adequate reduction and optimize acetabular coverage. The study's procedural protocols were developed in consultation with senior pediatric orthopedic surgeons experienced in both techniques and piloted to establish feasibility before patient enrollment commenced. In this manner, the investigation aims to refine the understanding of arthroscopic-assisted hip reconstruction in the pediatric population, providing insights that may influence future surgical guidelines, training curricula, and patient care pathways.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with DDH (Tönnis grade II-IV)
* Age range: 12 to 24 months at the time of the first surgical reduction
* A documented failed attempt at conservative reduction (e.g., closed reduction) prior to enrollment

Exclusion Criteria:

* Presence of neuromuscular disorders
* Teratologic hip dislocation
* Prior surgical intervention on the affected hip
* Incomplete radiographic documentation (missing radiographs at any of the required assessment intervals)

Ages: 1 Year to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
rate of hip redislocation documented clinically and radiographically at 6, 12, and 24 months postoperatively. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Erbil Teaching Hospital, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: No